CLINICAL TRIAL: NCT04418791
Title: Modified Intermittent Fasting in Psoriasis Trial: a Randomized Controlled Open Crossover Clinical Trial to Investigate the Effects of a Dietary Intervention on the Gut-skin Axis in Patients with Psoriasis
Brief Title: Modified Intermittent Fasting in Psoriasis
Acronym: MANGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BC-6977
Record Dates: First submitted 2019-12-18; First posted 2020-06-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Psoriasis Vulgaris; Psoriasis
Keywords: Psoriasis; Fasting; Modified intermittent fasting; Leaky gut; Intestinal barrier
MeSH Terms: conditions — Psoriasis; Fasting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Skin severity will be assessed by blinded physician for quantification of Psoriasis Area Severity Index (PASI) and Body Surface Area (BSA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MIF-regular (Experimental): MIF-regular will start with modified intermittent fasting. After 12 weeks, this arm will return to regular diet with no fasting intervention.
  Interventions: Behavioral: Modified Intermittent Fasting followed by Regular Diet
- Regular-MIF (Experimental): Regular-MIF will start with regular diet with no fasting. After 12 weeks, this arm will start with modified intermittent fasting.
  Interventions: Behavioral: Regular Diet followed by Modified Intermittent Fasting

INTERVENTIONS:
Behavioral: Modified Intermittent Fasting followed by Regular Diet — Modified intermittent fasting (MIF) means fasting for 2 non-consecutive days/week. Fasting is defined as consuming less than 500 kcalories in 1 day (in the course of max. 6 hours). After 12 weeks of fasting, a period of 12 weeks with a regular diet follows.
  Arms: MIF-regular
Behavioral: Regular Diet followed by Modified Intermittent Fasting — Regular diet means subject can eat as usual for 12 weeks. Next, a period of 12 weeks fasting follows: modified intermittent fasting (MIF) means fasting for 2 non-consecutive days/week. Fasting is defined as consuming less than 500 kcalories in 1 day (in the course of max. 6 hours).
  Arms: Regular-MIF

SUMMARY:
The complexity of psoriasis is partially affected by dietary effects, and some diets have shown to be beneficial in psoriasis. Intermittent fasting has been shown to improve many of these disturbances, even inflammatory parameters such as TNF and CRP. Individuals with psoriasis have been reported to have impaired intestinal integrity and it has been suggested that gut health affects skin health, pointing towards a gut-skin axis. Understanding how dietary lifestyles can affect epithelial lineages such as the skin and gut, will greatly improve our understanding on the development of psoriasis. Modified intermittent fasting (MIF) of 2 non-consecutive days has shown to have positive metabolic effects, yet its effect on gut and skin remains underexplored.

DETAILED DESCRIPTION:
To study the role of gut health, more specifically the intestinal barrier, in individuals with psoriasis and the effects of fasting on both organs in a prospective cohort cross-over study. The investigators will test whether MIF can improve (i) skin lesions (clinical and molecular level), (ii) intestinal integrity markers such as zonulin, IFABP and sCD14, and (iii) the timing of these improvements. As such, it can be determined whether fasting benefits psoriasis and gut health. MIF will consist of a limited calorie uptake of 500 kcal for 2 days a week. The remaining days of the week are as usual. Gut and skin health will be tested at the molecular level during 12 weeks with another crossover of 12 weeks (alternating between MIF and usual diet).

ELIGIBILITY:
Inclusion Criteria:

* Mild psoriasis (PASI < 10)
* At least BMI of 20
* Stable weight for last 3 months
* Topical treatment
* Availability of smartphone and willing to install app
* Willing to attend dematology clinic at Ghent University Hospital

Exclusion Criteria:

* Underweight and/or following strict diet
* Use of anti, pre and/or probiotics (last 3 months)
* Use of immunosuppressants (last 3 months)
* Smoking
* Consumption of fish oil
* Diagnosed diabetes (type ½)
* Excessive physical activity
* Pregnancy or breastfeeding
* More than 14 alcohol units/week
* History of cardiac condition(s)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-17 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Improvement in psoriasis severity amongst subjects during and after intervention defined as Psoriasis Area Severity Index | 12 and 26 weeks
  Change in Psoriasis Area Severity Index
Psoriasis severity amongst subjects during and after intervention defined as Body Surface Area | 12 and 26 weeks
  Change in Body Surface Area

SECONDARY OUTCOMES:
Total body fat during and after intervention to baseline | 12 and 26 weeks
  Change in total body fat
Weight during and after intervention to baseline | 12 and 26 weeks
  Change in weight (kg)
Body Mass Index during and after intervention to baseline | 12 and 26 weeks
  Change in Body Mass Index measured as weight (kg) and height (m) (kg/m^2)
Waist circumference during and after intervention to baseline | 12 and 26 weeks
  Change in waist circumference (cm)
Inflammation markers in serum during and after intervention to baseline | 12 and 26 weeks
  Change in serological markers for inflammation [pg/ml]
Inflammation markers in skin during and after intervention to baseline | 12 and 26 weeks
  Change in cutaneous markers for inflammation [pg/ml]
Metabolic markers in serum during and after intervention to baseline | 12 and 26 weeks
  Change in serological markers for metabolism [pg/ml]
Metabolic markers in skin during and after intervention to baseline | 12 and 26 weeks
  Change in cutaneous markers for metabolism [pg/ml]
Permeability markers in serum during and after intervention to baseline | 12 and 26 weeks
  Change in serological markers for permeability [pg/ml]
Permeability markers in feces during and after intervention to baseline | 12 and 26 weeks
  Change in fecal markers for permeability [pg/ml]
Visual Analogue Scale Satisfaction | 12 and 26 weeks
  Score of subject's rating of satisfaction and/or feasibility on intervention based on a Visual Analogue Scale going from 0 (not satisfied at all) to 10 (very satisfied)
Study completion by subjects | 12 and 26 weeks
  Number of subjects who completed the study successfully (adherence to intervention) as a percentage.
Quality of life during and after intervention to baseline | 12 and 26 weeks
  Change in Dermatology Life Quality Index (absolute and relative)
Prediction of dietary intake | 12 and 26 weeks
  Correlation of outcomes 1-15 in relation to dietary intake

CONTACTS AND LOCATIONS:
Overall Officials: Jo Lambert, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Department of Head & Skin, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grine L, Hilhorst N, Michels N, Abbeddou S, De Henauw S, Lambert J. The Effects of Modified Intermittent Fasting in Psoriasis (MANGO): Protocol for a Two-Arm Pilot Randomized Controlled Open Cross-over Study. JMIR Res Protoc. 2022 Feb 23;11(2):e26405. doi: 10.2196/26405. PMID 35195533
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35195533/